CLINICAL TRIAL: NCT06025799
Title: Effect of Mindfulness-based Stress Reduction Intervention on Psychological Distress and Hope Among Female Patients Undergoing Radiotherapy for Breast Cancer: A Randomized Control Trial
Brief Title: Effect of Mindfulness-based Stress Reduction Intervention on Psychological Distress and Hope Among Female Patients Undergoing Radiotherapy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Heba Mohamed Abdelaal, Assistant professor at Psychiatric& Mental Health Nursing, Faculty of Nursing, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00013620/8/2023
Record Dates: First submitted 2023-08-30; First posted 2023-09-06 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer Female
Keywords: Mindfulness-based stress reduction; Psychological Distress; Hope; Female patients; Radiotherapy; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Mindfulness-based stress reduction intervention" (Experimental): patients who will be under routine hospital care as well as Mindfulness-Based Stress Reduction (MBSR) program The Mindfulness-Based Stress Reduction (MBSR) program consists of eight sessions focusing on reducing stress and improving well-being. Participants learn and practice mindfulness techniques such as mindful eating, breathing, body scan, and meditation. The program emphasizes self-responsibility, developing coping strategies, and applying mindfulness daily. Participants engage in formal mindfulness practices, reflect on their experiences, and receive guidance on continuing their mindfulness journey after the program. The goal is to cultivate resilience, enhance well-being, and reduce stress.
  Interventions: Behavioral: Mindfulness-based stress reduction intervention
- " routine hospital care" (No Intervention): Female cancer patients who will be under routine hospital care

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction intervention — The Mindfulness-Based Stress Reduction (MBSR) program consists of eight sessions focusing on reducing stress and improving well-being. Participants learn and practice mindfulness techniques such as mindful eating, breathing, body scan, and meditation. The program emphasizes self-responsibility, developing coping strategies, and applying mindfulness daily. Participants engage in formal mindfulness practices, reflect on their experiences, and receive guidance on continuing their mindfulness journey after the program. The goal is to cultivate resilience, enhance well-being, and reduce stress.
  Arms: "Mindfulness-based stress reduction intervention"

SUMMARY:
Breast cancer is a significant issue in Egypt, affecting a large number of women and impacting their psychological well-being. Younger patients and those undergoing adjuvant therapy or radiotherapy are particularly susceptible to psychological distress. Psychological counseling and support groups can help improve patients' quality of life and social functioning. Hope plays a crucial role in the treatment process, as it is associated with positive outcomes and serves as a protective mechanism against stress and disease. Mindfulness-Based Stress Reduction (MBSR) is an intervention that can reduce stress and depression in cancer patients. It involves cultivating awareness of the present moment and has positive effects on quality of life. Investigating the impact of MBSR on psychological distress and hope in women undergoing radiotherapy for breast cancer is important for providing effective support during treatment.

The aim of this study is to:

Examine the effect of the Mindfulness-Based Stress reduction intervention on psychological distress and hope among female patients undergoing radiotherapy for breast cancer.

RESEARCH HYPOTHESIS Female patients undergoing radiotherapy for breast cancer who attend Mindfulness-Based Stress reduction intervention sessions exhibit higher levels of hope and lower levels of psychological distress compared to those who receive conventional hospital treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients with post-mastectomy (within one to six months).
* Able to communicate verbally.
* Able to read and write.
* Willing to participate in the study.

Exclusion Criteria:

* other associated diseases such as (renal disease, ischemic heart disease, liver disease) will e excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Adult female patients with post-mastectomy to decrease the confounding factors.
Enrollment: 100 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Five Factors Mindfulness Questionnaire (FFMQ) | 9 weeks
  The Baer et al. (2006) scale is a 39-item questionnaire designed to measure different aspects of mindfulness. It uses a five-point Likert scale, with responses ranging from 1 (never or very rarely true) to 5 (very often or always true). The scale consists of five subscales: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience.
  Observing subscale: Measures the tendency to notice or attend to internal and external phenomena.
  Describing subscale: Assesses the ability to label observed phenomena, such as thoughts and emotions.
  Acting with awareness subscale: Reflects the extent to which individuals engage with full awareness in their current experience or activity.
  Non-judging subscale: Assesses nonjudgmental awareness of current experience without evaluation.
  Non-reactivity subscale: Measures the ability to notice internal phenomena without reacting to them.
Depression Anxiety and Stress Scale 21 (DASS-21) | 9 weeks
  It is a self-reported scale developed by Lovibond, & Lovibond, (1995). The three subscales of the DASS 21 measure the negative emotional states of depression, anxiety, and stress (i.e., nervous tension and irritability, which are factorially distinct from depression and anxiety). Participants scored questions such as "I thought that as a person I wasn't worth much" (from "0" =did not apply to me at all to "3" =applied very much to me or most of the time). A total score out of 21 was determined for each subscale and then multiplied by 2 to be equivalent to the full-scale DASS scores. At least 10 (depression), 8 (anxiety), and 15 (stress) ratings indicated psychological distress levels for each item. Distress severity was categorized as mild, moderate, severe, and very severe.
The Herth Hope Index (HHI) | 9 weeks
  The Herth Hope Index (HHI) is a clinical-setting adaptation form of the Herth Hope Scale (HHS). This scale was developed by Herth, at Minnesota State in the USA (Herth, 1992). It is composed of 12 items, which are rated on a four points Likert scale. The responses ranged from 1 (strongly disagree) to 4 (strongly agree). Items 3 and 6 are reversed in their score. The twelve items are summed to obtain a total score that ranges from 12 to 48, with a higher score equating to a higher level of hope. The instrument contains three factors, namely temporality & future, positive readiness & expectancy, and finally interconnectedness with self and others.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carlson LE, Ursuliak Z, Goodey E, Angen M, Speca M. The effects of a mindfulness meditation-based stress reduction program on mood and symptoms of stress in cancer outpatients: 6-month follow-up. Support Care Cancer. 2001 Mar;9(2):112-23. doi: 10.1007/s005200000206. PMID 11305069